CLINICAL TRIAL: NCT01818557
Title: Frequency of Blood Glucose Monitoring in Patients With Gestational Diabetes: A Randomized, Non-Inferiority Pilot Study
Brief Title: Frequency of Blood Glucose Monitoring in Patients With Gestational Diabetes
Acronym: GLIMPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-13-0719
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Gestational Diabetes
Keywords: glucose monitoring; gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Every day blood glucose testing (No Intervention): Patients will test their blood glucose values 4 times every day
- Every other day blood glucose testing (Experimental): Patients will test their blood glucose 4 times every other day
  Interventions: Behavioral: Blood glucose testing

INTERVENTIONS:
Behavioral: Blood glucose testing — Patients will be assigned either to blood glucose monitoring done every day (during a fasting state and 2 hours after breakfast, lunch and dinner) continued throughout gestation or to blood glucose monitoring done every other day with the same timeframes outlined above.
  Arms: Every other day blood glucose testing

SUMMARY:
The incidence of gestational diabetes mellitus (GDM) is increasing. GDM requires patients to test their blood glucose at least four times daily. The investigators propose to prospectively evaluate blood glucose testing done every day compared to every other day. The primary goal is to establish the most cost-effective modality while still being able to detect patients who require therapy in a timely fashion. The investigators plan to evaluate this new management scheme utilizing a non-inferiority trial design.

The investigators primary research question is the following: When managing patients with GDM, is every other day blood glucose testing non-inferior compared to every day blood glucose testing, as measured by the difference of less than 5% in birth weight?

DETAILED DESCRIPTION:
This study is a prospective randomized, non-inferiority clinical trial of pregnant women diagnosed with gestational diabetes. Patients with GDM diagnosed between 20 weeks 0 days and 32 weeks 0 days of gestation will be recruited. Diagnosis of GDM will be based on Carpenter and Coustan criteria for an abnormal 3-hr 100 gram oral glucose tolerance test, as currently supported by the American College of Obstetricians and Gynecologists (ACOG). Patients whose 1-hr, 50 gram oral glucose challenge test exceeds 200 mg/dl will not require a 3-hr oral glucose tolerance test (OGTT). If the patient meets the inclusion and exclusion criteria listed below, she will be offered participation in the trial and randomized to every day blood glucose testing or every other day blood glucose testing for the remainder of her pregnancy.

After the diagnosis of GDM, and before recruitment to the study, all patients will be provided counseling and education and will attempt adequate blood glucose control with medical nutritional therapy alone for one week. During this period, all patients will test their blood glucose values daily. Only after this week is completed will a subject be approached for participation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 20 weeks 0 days and 32 weeks 0 days of gestation.
* Singleton pregnancies
* Maternal age over 18 years
* Patients able to read and write in English or Spanish,
* Diagnosis of gestational diabetes mellitus using criteria supported by the American College of Obstetrics and Gynecology (ACOG).
* Patients identified as not requiring medical therapy (insulin or glyburide) after the first week of initial blood glucose monitoring.

Exclusion Criteria:

* Diagnosis of GDM made by any method or criteria other than the one outlined above
* Women with pre-existing diabetes mellitus
* Patients under the age of 18 years
* Patients known to be carrying a fetus with a fetal anomaly that requires either prenatal or postnatal surgery, requires early delivery or is at risk for intrauterine growth restriction (IUGR)
* Patients carrying multiple gestations
* Patients with past history of gastric bypass
* Patients with poorly controlled asthma, defined as the need for oral/inhaled corticosteroids to control symptoms
* Patients with chronic hypertension requiring medical therapy
* Patients currently on methadone/suboxone therapy
* Patients currently on any steroid therapy, regardless of the dose or route of administration
* Patients demonstrating poor compliance during the first week of initial blood glucose monitoring, defined as <20% of expected values actually recorded during the one-week period of initial monitoring

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Neonatal weight | At birth
  In patients with GDM, every other day blood glucose testing is non-inferior to every day blood glucose testing, as measured by the difference of less than 5% in birth weight

SECONDARY OUTCOMES:
Macrosomia | At birth
  To determine if every other day testing is associated with a greater rate of macrosomia, defined as birth weight > 4,000 grams, than every day blood glucose testing

CONTACTS AND LOCATIONS:
Overall Officials: Hector Mendez-Figueroa, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - Geisinger Health System, Danville, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - The University of Texas Health Science Center, Houston, Houston, Texas

REFERENCES:
- [Derived] Mendez-Figueroa H, Schuster M, Maggio L, Pedroza C, Chauhan SP, Paglia MJ. Gestational Diabetes Mellitus and Frequency of Blood Glucose Monitoring: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):163-170. doi: 10.1097/AOG.0000000000002101. PMID 28594772